CLINICAL TRIAL: NCT02037113
Title: Outcomes of Femoro-popliteal Disease After Stent Deployment Under Intravascular Ultrasound Guidance (CRI14-007)
Brief Title: Outcomes of Femoro-popliteal Disease After Stent Deployment Under Intravascular Ultrasound Guidance
Acronym: IVUS-PAD
Status: Terminated | Type: Observational
Why Stopped: PI left institution--only 8 subjects were enrolled.
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L14-047
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Peripheral Arterial Disease
Keywords: IVUS; PAD; Femoro-popliteal disease; Intravascular ultrasound
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient underwent PAD-Stent: Patient who underwent angioplasty and/or atherectomy with stent placement for Femoro-popliteal disease and Intravascular ultrasound was performed after stent deployment.

SUMMARY:
This is a prospective, single-center study. The patients with peripheral arterial disease who underwent abdominal aortograms with runoff (which are arteriograms of the lower abdominal aorta and arteries in the legs) and Intravascular Ultrasound after stent deployment will be enrolled in the study. All patients who participated in the study will be treated according to standard of care.

HYPOTHESIS The higher degree of plaque burden on landing zone has an effect on restenosis on peripheral artery intervention.

SPECIFIC AIMS

1. To determine intravascular ultrasound parameters of stent deployment and outcomes of Femoro-popliteal Disease
2. To determine clinical risk factors and outcomes of Femoro-popliteal Disease
3. To obtain data that will eventually support development of a predictive model for ISR in Femoro-popliteal Disease

METHODOLOGY Visit 1: After consent is given

The subject will receive standard follow-up care. A member of the research team will collect information such as the subject's age, sex, ethnicity, and medical information from the subject's medical record.

Visits 2-5: 1 day after enrollment, and at months 3 (+- 2 weeks), 6 (+- 2 weeks), and 12 (+- 2 weeks)

The subject will complete standard follow-up appointment at TTUHSC. This may include a Doppler ultrasound.

A member of the research team will record information such as medications, ultrasounds, and need for additional care related to the subject's stent.

The subject will complete the questionnaire on leg pain and mobility.

DETAILED DESCRIPTION:
SUBJECT POPULATION:

- The patients who have peripheral arterial disease and underwent elective abdominal aortograms with runoff with peripheral artery intervention in University Medical Center hospital, Lubbock Texas, during January 2014 to December 30, 2015.

INCLUSION CRITERIA:

* 25-89 years of age
* Admitted for elective abdominal aortograms with runoff.
* Underwent Angioplasty and/or atherectomy with stent placement for Femoro-popliteal disease.
* Intravascular ultrasound was performed after stent deployment.

EXCLUSION CRITERIA:

* Patients who had prior Femoro-popliteal artery surgery or bypass in the same limb.
* Stent placement for lesions above inguinal ligament or below popliteal artery.
* The patient who presented with acute limb ischemia.
* Unable to follow-up in TTUHSC clinic.

ELIGIBILITY:
Inclusion Criteria:

* 25-89 years of age
* Admitted for elective abdominal aortograms with runoff.
* Underwent Angioplasty and/or atherectomy with stent placement for Femoro-popliteal disease.
* Intravascular ultrasound was performed after stent deployment.

Exclusion Criteria:

* Patients who had prior Femoro-popliteal artery surgery or bypass in the same limb.
* Stent placement for lesions above inguinal ligament or below popliteal artery.
* The patient who presented with acute limb ischemia.
* Unable to follow-up in TTUHSC clinic.

Ages: 25 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who have peripheral arterial disease and underwent elective abdominal aortograms with runoff with peripheral artery intervention in University Medical Center hospital, Lubbock Texas, during January 2014 to December 30, 2015.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
In Stent Restenosis | 1 years
Redo procedure | 1 year
Early and late stent thrombosis | 1 year
Acute ischemic event | 1 year

SECONDARY OUTCOMES:
All causes mortality | 1 year
  to be obtained from UMC Cath-Lab NCDR registry

CONTACTS AND LOCATIONS:
Overall Officials: Alex Suarez, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sigwart U, Puel J, Mirkovitch V, Joffre F, Kappenberger L. Intravascular stents to prevent occlusion and restenosis after transluminal angioplasty. N Engl J Med. 1987 Mar 19;316(12):701-6. doi: 10.1056/NEJM198703193161201. PMID 2950322
- [Background] Conte MS, Bandyk DF, Clowes AW, Moneta GL, Seely L, Lorenz TJ, Namini H, Hamdan AD, Roddy SP, Belkin M, Berceli SA, DeMasi RJ, Samson RH, Berman SS; PREVENT III Investigators. Results of PREVENT III: a multicenter, randomized trial of edifoligide for the prevention of vein graft failure in lower extremity bypass surgery. J Vasc Surg. 2006 Apr;43(4):742-751; discussion 751. doi: 10.1016/j.jvs.2005.12.058. PMID 16616230
- [Background] Reifsnyder T, Grossman JP, Leers SA. Limb loss after lower extremity bypass. Am J Surg. 1997 Aug;174(2):149-51. doi: 10.1016/s0002-9610(97)90074-x. PMID 9293832
- [Background] Sullivan TM, Childs MB, Bacharach JM, Gray BH, Piedmonte MR. Percutaneous transluminal angioplasty and primary stenting of the iliac arteries in 288 patients. J Vasc Surg. 1997 May;25(5):829-38; discussion 838-9. doi: 10.1016/s0741-5214(97)70212-x. PMID 9152310
- [Background] Martinez R, Rodriguez-Lopez J, Diethrich EB. Stenting for abdominal aortic occlusive disease. Long-term results. Tex Heart Inst J. 1997;24(1):15-22. PMID 9068134
- [Background] Leon LR Jr, Dieter RS, Gadd CL, Ranellone E, Mills JL Sr, Montero-Baker MF, Gruessner AC, Pacanowski JP Jr. Preliminary results of the initial United States experience with the Supera woven nitinol stent in the popliteal artery. J Vasc Surg. 2013 Apr;57(4):1014-22. doi: 10.1016/j.jvs.2012.10.093. PMID 23535039
- [Background] Schillinger M, Sabeti S, Loewe C, Dick P, Amighi J, Mlekusch W, Schlager O, Cejna M, Lammer J, Minar E. Balloon angioplasty versus implantation of nitinol stents in the superficial femoral artery. N Engl J Med. 2006 May 4;354(18):1879-88. doi: 10.1056/NEJMoa051303. PMID 16672699